CLINICAL TRIAL: NCT04996277
Title: A Prospective Evaluation of Clinical Impact of Physiology Versus Optical Coherence Tomography Guided PCI in STEMI Patients Without Undergoing Primary PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CCRF Inc., Beijing, China (Industry)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Yaling Han, M.d., Ph.D., Academician/chief physician, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OCT-STEMI-2020
Record Dates: First submitted 2021-07-23; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Cerebral Angiography; Thrombolytic Therapy

STUDY DESIGN:
Intervention Model Description: In this study, 300 subjects with target vessel stenosis of 50%-90% confirmed to be suitable for stent implantation by angiographic evaluation will be recruited and randomly assigned to FFR, OCT or Angio group according to 1:1:1. FFR group: Patients with FFR ≤0.8 were treated with PCI; FFR > 0.8 patients will receive drug therapy; All patients will undergo OCT examination. OCT group: if MLA< 4.5mm2 patients will receive PCI; Other patients will be treated with medication; All patients will be examined for FFR. Angio group: The appropriate treatment (stent implantation) will be given according to the evaluation of the doctor.
Masking Description: During the study, it is difficult for researchers, operators and patients to blind the method due to objective reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fractional Flow Reserve (Experimental): Patients with FFR ≤ 0.8 will undergo PCI Patients with FFR > 0.8 will be treated with medication For study purposes, all patients will undergo OCT (subject's treatment strategy will be based on FFR results, e.g., stent-implanted OCT).
  Interventions: Procedure: angiography; Procedure: Thrombus suction; Procedure: Fibrinolytic therapy; Behavioral: Medication stabilized the condition
- Optical CoherenceTomography (Experimental): Patients with MLA < 4.5mm² will undergo PCI Other patients will be treated with medication For study purposes, all patients will undergo FFR (subject's treatment strategy is based on OCT results; reference to FFR results is not recommended)
  Interventions: Procedure: angiography; Procedure: Thrombus suction; Procedure: Fibrinolytic therapy; Behavioral: Medication stabilized the condition
- angiography (Experimental): Appropriate treatment (implantation of stents) will be given according to the evaluation of the physician.
  Interventions: Procedure: angiography; Procedure: Thrombus suction; Procedure: Fibrinolytic therapy; Behavioral: Medication stabilized the condition

INTERVENTIONS:
Procedure: angiography — All STEMI patients will be treated according to the hospital's standard procedures and the plaque will be monitored for 7-30 days to stabilize. Treatment options for STEMI include: March thrombus aspiration without balloon or stent implantation; Stabilization with drug therapy in a relatively small hospital that does not provide PCI, and transfer to a tertiary hospital for further evaluation; Thrombolytic therapy.
Procedure: Thrombus suction — All STEMI patients will be treated according to the hospital's standard procedures and the plaque will be monitored for 7-30 days to stabilize. Treatment options for STEMI include: March thrombus aspiration without balloon or stent implantation; Stabilization with drug therapy in a relatively small hospital that does not provide PCI, and transfer to a tertiary hospital for further evaluation; Thrombolytic therapy.
Procedure: Fibrinolytic therapy — All STEMI patients will be treated according to the hospital's standard procedures and the plaque will be monitored for 7-30 days to stabilize. Treatment options for STEMI include: March thrombus aspiration without balloon or stent implantation; Stabilization with drug therapy in a relatively small hospital that does not provide PCI, and transfer to a tertiary hospital for further evaluation; Thrombolytic therapy.
Behavioral: Medication stabilized the condition — All STEMI patients will be treated according to the hospital's standard procedures and the plaque will be monitored for 7-30 days to stabilize. Treatment options for STEMI include: March thrombus aspiration without balloon or stent implantation; Stabilization with drug therapy in a relatively small hospital that does not provide PCI, and transfer to a tertiary hospital for further evaluation; Thrombolytic therapy.

SUMMARY:
This study of physiologically functional FFR in STEMI patients without direct PCI treatment will provide unique data on plaque progression and risk factors.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multicenter clinical study that plans to continuously enroll patients with STEMI who, for various reasons, have not received direct PCI treatment within 48 hours of symptom onset. All STEMI patients will be treated according to the hospital's standard procedures and will continue to watch for plaque stability for 7 to 30 days. Treatment options for STEMI include: progressive thrombus aspiration without balloon or stent implantation; Stabilization with medication in a relatively small hospital that could not provide PCI treatment and then transfer to a tertiary hospital for further evaluation; Thrombolytic therapy. After that, all patients underwent an angiogram to identify any residual stenosis in the culprit's blood vessels.

In this study, 300 subjects with target vessel stenosis of 50%-90% confirmed to be suitable for stent implantation by angiographic evaluation will be recruited and randomly assigned to FFR, OCT or Angio group according to 1:1:1. FFR group: Patients with FFR ≤0.8 were treated with PCI; FFR > 0.8 patients will receive drug therapy; All patients will undergo OCT examination. OCT group: if MLA< 4.5mm2 patients will receive PCI; Other patients will be treated with medication; All patients will be examined for FFR. Angio group: The appropriate treatment (stent implantation) will be given according to the evaluation of the doctor.

All patients were followed up at 1 month (±7d), 6 months (±14d) and 12 months (±30d) after surgery, respectively. Target lesion failure (TLF), including cardiogenic death, target vessel myocardial infarction (TV-MI), or clinically indicated target lesion revascularization (TLR), was used as the primary end point. Secondary end points included the incidence of major adverse cardiovascular events (MACE) at 1 year postoperatively. The clinical composite end points included: All due to death, Arc-defined stent thrombotic events, non-fatal myocardial infarction, clinically driven target vessel revascularization, or readmission due to unstable angina pectoris or aggravation of angina; Patients in the FFR group and OCT group were treated with a change of treatment strategy (pre-PCI: change of stent implantation strategy; After PCI: with or without additional intervention).

Each research center shall operate and test in accordance with the operating procedures uniformly described in the scheme to ensure the consistency of the test operation.

Clinical event committee (CEC) : a clinical event committee will be composed of independent cardiologists not involved in this study to reevaluate all reported deaths, myocardial infarction, revascularization, and thrombotic events.

A total of 300 STEMI patients who did not receive direct PCI treatment within 48 hours after symptom onset due to different reasons are planned to be enrolled in 16 centers nationwide. The overall study time is about 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. age ≤ 18 ≤75;
2. 7-30 days after onset of STEMI;
3. PCI was not performed for the following reasons:

   1. Stabilize the condition at a hospital that is unable to provide PCI and then refer to a tertiary hospital for further evaluation;
   2. Previous emergency angiography without balloon dilatation or stent implantation; Emergency thrombus aspiration without balloon dilation or stent placement;
4. Patients with target lesion stenosis of 50%-90%, GRADE 3 TIMI blood flow and indications for stent implantation after receiving STEMI treatment in accordance with hospital standard procedures.

Exclusion Criteria:

1. Left main disease or bypass disease;
2. Intolerance to research drugs, metal alloys or contrast agents;
3. Life expectancy is less than a year;
4. PCI was performed on previous target vessels;
5. Previous coronary artery bypass grafting;
6. cardiogenic shock or LVEF< 35%;
7. Severe renal or liver dysfunction;
8. Hemodynamic instability;
9. The degree of pathological stenosis of criminals was > 90% or < 50%;
10. Target vessel TIMI blood flow ≤ grade 2;
11. A surgical plan within 6 months after the initial operation;
12. Had clinical indications of intolerance to 12-month DAPT therapy;
13. Unable to provide written proof of informed consent;
14. Patients who were enrolled in other clinical trials at the time of enrollment and did not meet the primary study endpoint.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 1 year after baseline surgery
  These include cardiogenic death, target vascular-associated myocardial infarction, and ischaemic driven revascularization of target lesions

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 1 year after baseline surgery
  All-cause death; ARC defined stent thrombosis events; This is a nonfatal myocardial infarction Anyway, a clinically-driven revascularization of a target blood vessel or hospital re-admission due to unstable angina or worsening angina
Incidence of changes in treatment strategy in FFR and OCT patients | 1 year after baseline surgery
  Change of stent implantation strategy before PCI and additional intervention or no additional intervention after PCI